CLINICAL TRIAL: NCT05595694
Title: Incidence and Duration of Acute Kidney Injury After Elective Total Joint Arthroplasty With The Use of Perioperative Celecoxib as One of the Multimodal Analgesia Regime: A Retrospective Case Control Study
Brief Title: Acute Kidney Injury After Elective Total Joint Arthroplasty
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Honorary Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW22-230
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a retrospective review of 1320 patients in our database who underwent elective primary and revision TJA in Queen Mary Hospital, Hong Kong from from January 2018 to December 2021. No intervention was involved.

SUMMARY:
Total joint arthroplasty (TJA) is a common orthopedic procedure to treat patients with end-stage knee arthritis. Over 4,000 TJA were performed in the Hong Kong public hospitals in the past 12 months (July 2020 - June 2021) and the demand for this procedure is ever increasing with time. TJA are rehabilitative surgeries with an aim to accelerate patient ambulation and minimize hospital stay. To facilitate this process, multi-disciplinary enhanced recovery after surgery (ERAS) programs are implemented. This involves surgeons, anaesthetists, physiotherapists and nurses who follow an integrated care pathway to allow early patient mobilization and hospital discharge. The program reduces the hospital length of stay and this can reduce the risk of complications and mortality. One of the major challenges in TJA is postoperative pain. TJA is a very painful procedure with up to 50% of patients have moderate to severe pain (numeric rating scale >4) immediately after surgery. This can delay patient mobilization and hinder postoperative recovery. Severe postoperative pain is also associated with an increased risk of infection, myocardial ischaemia, respiratory complications and the development of chronic pain. Therefore, an effective multimodal analgesia is an essential component in the ERAS program. It combines different oral analgesics to limit opioid use and its related side effects. Celecoxib has been shown to reduce pain and opioid use after TJA. It is therefore recommended to be used routinely. However, its potential nephrotoxic property has led to its judicious use, especially in patients with preoperative chronic renal failure. Postoperative acute kidney injury (AKI) is an independent risk factor for mortality, cardiovascular complications and hospital length of stay6. However, the studies assessing the incidence of AKI following TJA are scarce, and with conflicting results.

Therefore, the aim of our study is to retrospectively review the incidence and duration of AKI following elective TJA in a tertiary institution. We will evaluate the effect of celecoxib in our multimodal analgesia regimen on the risk of postoperative AKI and determine the risk factors associated.

ELIGIBILITY:
Inclusion Criteria:

* Patients data in our database who underwent elective primary and revision TJA in Queen Mary Hospital, Hong Kong from from January 2018 to December 2021.

Exclusion Criteria:

* Patients with rheumatoid arthritis.
* Missing of essential data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent elective primary and revision TJA in Queen Mary Hospital, Hong Kong from from January 2018 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1077 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | From postoperative day 0 to day 5
  Daily serum creatinine level from postoperative day 0 up to day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No